CLINICAL TRIAL: NCT04012385
Title: An Intervention Model for the Prevention of Infertility in Healthy Young Men Living in Highly Polluted Areas
Brief Title: Effects of Lifestyle Changes on Semen Quality in Healthy Young Men Living in Highly Polluted Areas (FAST)
Acronym: FAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Sanitaria Locale Salerno (Other)
Collaborators: Istituto clinico Città di Brescia (Unknown); Università degli Studi di Brescia (Other); Istituto Superiore di Sanità (Other); Ministero della Salute, Italy (Other); ISA-CNR, Avellino (Unknown); Molecular Epidemiology and Environmental Epigenetics Lab (Unknown)
Responsible Party: Principal Investigator, LUIGI MONTANO, Principal Investigator, Azienda Sanitaria Locale Salerno
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: J59D1600132001
Record Dates: First submitted 2019-02-15; First posted 2019-07-09 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Fertility Disorders
Keywords: Lifestyle; Fertility; Nutrition; Environmental Pollution

STUDY DESIGN:
Intervention Model Description: Primary purpose of the study is the improvement of semen quality in healthy young men living in highly polluted areas, operating on two specific lifestyle factors, that are nutrition and physical activity. Overall, 450 subjects will be enrolled (150 for single recruiting area) and they will be assigned by chance to one of the two arms of the study, named "Control group" and "Intervention group". Every subject is identified by means of an individual alphanumeric code that does not specifies which group they belong to, in order to mask to all the outcomes assessors the membership to one arm or another.
Who Masked: Outcomes Assessor
Masking Description: A specific alphanumeric code is assigned to each participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Subjects assigned to control group receives only a booklet including the recommendations for a correct diet by the Italian National Institute for Research on Food and Nutrition (INRAN), presently called (CRA-NUT) .
- Intervention (Experimental): Subjects assigned to the intervention group will follow a nutritional pathway based on a Mediterranean diet pattern for 4 months and receive suggestions on the regular practice of physical activity, under the guide of some nutritionists, who will propose individualized diets for each subject.
  All subjects of both groups will undergo urologic examination, measurement of weight, height and abdominal circumference, an interview on demographic data and lifestyle variables, and will provide blood and semen samples in fasting conditions, at the enrollment (baseline), at the end of the intervention phase (after 4 months) and at the end of follow-up (after 8 months).
  Interventions: Behavioral: lifestyle counseling

INTERVENTIONS:
Behavioral: lifestyle counseling — Nutritional plan and Physical activity goals
  Arms: Intervention

SUMMARY:
We planned a randomized controlled trial (RCT) with the main aim to evaluate the effects of lifestyle changes on semen quality in healthy young men living in polluted areas in Italy. Secondary aims are to assess: a) the association between semen quality and biomarkers of early damage or inflammation; b) the associations between biomarkers of exposure to heavy metals and semen quality and biomarkers of early damage or inflammation; c) the associations between diet and physical activity and semen quality and biomarkers of early damage or inflammation; d) the effects of lifestyle changes on the blood and semen levels of heavy metals.

The RCT includes 450 young men living in one of the following three polluted areas:

1. a polychlorinated biphenyls (PCBs) polluted area in Brescia province, Lombardy region;
2. the valley of the Sacco river, with high levels of beta-hexachlorocyclohexane (β-HCH) originated by toxic waste dumps of industrial origin.
3. the "Land of Fires" in the Campania region, with a high concentration of illegal waste dumping and uncontrolled burning near cultivated fields.

Inclusion criteria are: a) healthy males aged 18- 22 years; b) residents in the area since at least 5 years; c) non smokers; d) non alcohol or drug users; e) normo-weight (18.5< BMI<24.99); f) no occupationally exposed to fertility toxics; g) not affected by chronic diseases. Subjects will be randomly assigned to an intervention or control group. The intervention group will follow a nutritional pathway and receive suggestions on practice of physical activity for 4 months, under the guide of some nutritionists, who will establish individualized diets for each subject. The control group will receive only a booklet including the dietary recommendations by the Italian National Institute for Research on Food and Nutrition. All subjects will undergo urologic examination, measurement of weight, height and abdominal circumference, an interview on demographic data, lifestyle variables, dietary habits, adherence to Mediterranean diet and physical activity, and will provide blood and semen samples in fasting conditions, at the enrollment (baseline), at the end of the intervention phase (after 4 months) and at the end of follow-up (after 8 months).

Laboratory analyses include the following:

* hematological parameters;
* semen quality parameters;
* prostate-specific antigen (PSA) in blood and semen;
* RedOx status parameters in semen;
* epigenetic analyses (DNA methylation) in blood lymphocytes and spermatozoa;
* content of heavy metals in blood and semen. The project has been approved by the local Ethics Committees. Differences of means and proportions of all variables between the intervention and control group and the associations between diet, physical activity and sperm and blood parameters will be assessed using common statistical tests for comparisons of means and proportions as a first step.

DETAILED DESCRIPTION:
Human semen quality is affected by genetic, metabolic, lifestyle and environmental factors. It is a sensitive marker of the general health status of an individual and a predictor of disease occurrence and mortality. Some studies suggested that a diet rich in anti-oxidant compounds and regular physical activity could improve semen quality. We planned a randomized controlled trial (RCT) with the main aim to evaluate the effects of lifestyle changes on semen quality in healthy young men living in three polluted areas in North, Centre and South Italy. Secondary aims are to assess: a) the association between semen quality and biomarkers of early damage or inflammation (prostate-specific antigen, RedOx status, epigenetic changes); b) the associations between biomarkers of exposure to toxic agents (heavy metals) and semen quality and biomarkers of early damage or inflammation; c) the associations between diet and physical activity and semen quality and biomarkers of early damage or inflammation; d) the effects of lifestyle changes on the blood and semen levels of heavy metals.

This RCT includes 450 healthy young men, aged 18-22 years, living in one of the following three polluted areas:

1. a polychlorinated biphenyls (PCBs) polluted area in Brescia province, Lombardy region;
2. the valley of the Sacco river, with high levels of beta-hexachlorocyclohexane (β-HCH) originated by toxic waste dumps of industrial origin.
3. the "Land of Fires" in the Campania region, with a high concentration of illegal waste dumping and uncontrolled burning near cultivated fields.

According to a 1:1 randomization plan, the young men will be assigned to an intervention or control group.

The subjects will be enrolled among high school and university students, after a 20 minute meeting with students in each class, during a lesson, and in the presence of the teacher, for explaining the study design and inviting them to participate. After a short self-administered screening questionnaire for excluding subject not suitable to the research, the potential candidates are invited to undergo a urologic visit, in a Urology and Fertility Unit, including a clinical examination and spermiogram analysis. In the same time, participant undergo a fasting blood sample for the analysis of common parameters (glycemia, cholesterolemia, ecc.), and measures of height, weight and abdominal circumference by trained dieticians. Then each dietician evaluated each participant's dietary habits and physical activity using the European Prospective Investigation into Cancer (EPIC) and nutrition questionnaire, the PREvención con DIeta MEDiterránea (PREDIMED), and the International Physical Activity Questionnaire (IPAQ).

Each urological visit, blood and semen sampling will be repeated with the same methodology in both intervention and control groups, at time 0 (baseline, enrollment), after 4 months (end of the intervention) and after 8 months (end of follow-up).

The intervention for changing lifestyle in the experimental group has been planned on the basis of previous experience of educational intervention in nutritional epidemiology. It should be noted that the Mediterranean diet is the focus of the intervention and that the aim of the intervention is not to loss weight but to increase the amount of anti-oxidants and anti-inflammatory dietary compounds. It is well known that also motivated subjects have difficulties in changing dietary habits. Therefore the change will be based on the following points: personalized diet (according to taste and practical reasons), progressive change (one objective a time), frequent contacts with dieticians (weekly contacts in the first month). The subjects are also invited to share dieticians' indications with their parents and especially the person who usually cooks at home. The dietician intervention has been planned with the help of Dr. Stefania Ubaldi, President of the European Lifestyle Medicine Organization (ELMO), Geneva.

The subjects included in the control group will receive only a booklet with present recommendations for Mediterranean diet at the enrollment (baseline), and will further contact only after 4 and 8 months.

Blood and semen samples will be collected and stored at -80° according to a standard protocol up to the time of laboratory analysis. Laboratory analyses include the following:

1. hematological parameters (whole blood count, glycemia, cholesterolemia, etc.);
2. semen quality parameters, according to the 2010 World Health Organization (WHO) criteria;
3. total and free prostate-specific antigen (PSA) in blood and semen;
4. RedOx status parameters in semen;
5. epigenetic analyses (DNA methylation) in blood lymphocytes and spermatozoa;
6. ICP-MS (Inductively Coupled Plasma Mass Spectrometry) analyses of heavy metals - aluminum (Al), antimony (Sb), arsenic (As), barium (Ba), beryllium (Be), cadmium (Cd), calcium (Ca), chromium (Cr), cobalt (Co), cuprum (Cu), iron (Fe), lead (Pb), lithium (Li) magnesium (Mg), manganese (Mn), molybdenum (Mo), nickel (Ni), potassium (K), selenium (Se), sodium (Na), strontium (Sr) and zinc (Zn) in blood and semen.

Differences of means and proportions of all variables between the intervention and control group and the associations between diet, physical activity and sperm and blood parameters will be assessed using common statistical tests for comparisons of means and proportions as a first step. Multivariable models, including multi-factor analysis of variance, multiple regression and multiple logistic regression, will then be used for assessing the associations when taking account of possible confounders. All the statistical tests are two-sided with p=0.05 as the threshold for refusal of the null hypothesis.

The two Urology and Fertility Units: a) Unità Operativa Complessa di Urologia, Ospedale S. Francesco d'Assisi di Oliveto Citra (SA), Azienda Sanitaria Locale (ASL) Salerno and b) the Unit of Hygiene, epidemiology and biostatistics and Unit of Urology of the University of Brescia will provide routine hematological parameters (whole blood count, glycemia, cholesterolemia, etc.) and semen quality parameters, according to the 2010 WHO criteria.

Each recruitment unit will collect and treat the biological samples, which will be sent to the laboratories for the specific analysis:

* Italian National Institute of Health, Rome: prostate-specific antigen in seminal plasma and in blood serum;
* Institute of Food Sciences, Italian National Research Council (ISA-CNR) of Avellino: RedOx status parameters in semen and ICP-MS analyses of heavy metals
* Epidemiology, Epigenetics And Toxicology (Epiget) Group of the University of Milan and Laboratory Biosafety and Risk Assessment of the Italian National Agency for New Technologies, Energy and Sustainable Economic Development (SSPT-TECS-BIORISC CR ENEA Casaccia): epigenetic analyses (DNA methylation) in blood lymphocytes and spermatozoa, respectively.

The data management and statistical analysis will be performed by the Unit of Hygiene, epidemiology and biostatistics of the University of Brescia.

ELIGIBILITY:
Inclusion Criteria:

* Young healthy men aged 18-22 years, who have been living at least for 5 years in one of the recruitment areas (Lombardy Region, "Land of fires" or Valley of the Sacco river)
* Normal weight (18,5 ≤ Body Mass Index < 25)
* Waist circumference < 102cm
* Having a normal sperm count (not azoospermic or cryptospermic)
* Drinking less than 5 alcohol units a week (1AU=125ml)
* Smoking less than 5 cigarettes (including e-cigarette, cigar, pipe)
* Smoking marijuana less than 3 times a month
* Must not have undergone urogenital surgery.
* Must not have suffered cancer disease and/or undergone chemo/radiotherapy.

Exclusion Criteria:

* Smoking more than 5 cigarettes a week
* Smoking marijuana more than 3 times a month
* Using drugs (other than marijuana)
* Drinking more than 5 alcohol units a week (1AU=125ml)
* Using dietary supplements (any type)
* Having a prior urogenital surgery (for varicocele: up to 12 months before the enrollment)
* Having suffered cancer and/or undergone chemo/radiotherapy
* Using anti-inflammatory drug on a regular basis (such as cortisone and/or NSAIDs) and/or having taken one of those drugs up to 72 hours before the collection of blood and semen samples.
* Using phosphodiesterase type 5 inhibitors (PDE5 inhibitor) up to 72 hours before the collection of blood and semen samples.
* Using steroids and/or anabolic hormones.
* Using dietary supplements and/or substances containing vegetal/animal extracts and/or trace elements up to 6 months before the enrollment.
* Fever status and/or antibiotic therapy up to 2 weeks before the enrollment.

Ages: 18 Years to 22 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Gender-based eligibility is directly related to the main purpose of the study, that is to evaluate the effects of lifestyle changes on male germ cells
Enrollment: 363 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-11-06 (Actual)

PRIMARY OUTCOMES:
changes in spermatozoa motility | assessed at baseline, after 4 and 8 months
  % total motility of spermatozoa
changes in Total Antioxidant Capacity (TAC) | assessed at baseline, after 4 and 8 months
  Total Antioxidant Capacity, measured in semen samples (mM)

SECONDARY OUTCOMES:
Sperm count | assessed at baseline, after 4 and 8 months from the enrollment
  millions of spermatozoa/ml sample
PSA | assessed at baseline and after 4 months from the enrollment
  Prostate-Specific Antigen in seminal plasma and in blood serum, measured in ng/ml
epigenetic analyses | assessed at baseline and after 4 months from the enrollment
  DNA-methylation status of Alu and L1 sequences
Trace elements | assessed at baseline and after 4 months from the enrollment
  dosage of trace elements in seminal plasma, semen and blood serum

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Montano, Dr, Principal Investigator — Urology Unit, "S. Francesco d'Assisi" Hospital, Oliveto Citra, A.S.L. Salerno
Locations (4):
- Italy (4):
  - Urology Unit "S. Francesco d'Assisi" Hospital, Oliveto Citra, Salerno
  - Unit of Hygiene, Epidemiology and Public Health, University of Brescia, Brescia
  - Unit of Urology - Istituto Clinico Città di Brescia, Brescia
  - Dpt. of Food safety, nutrition and veterinary public health, Italian National Institute of Health (ISS), Roma

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Stuppia L, Franzago M, Ballerini P, Gatta V, Antonucci I. Epigenetics and male reproduction: the consequences of paternal lifestyle on fertility, embryo development, and children lifetime health. Clin Epigenetics. 2015 Nov 11;7:120. doi: 10.1186/s13148-015-0155-4. eCollection 2015. PMID 26566402
- [Background] Vecoli C, Montano L, Andreassi MG. Environmental pollutants: genetic damage and epigenetic changes in male germ cells. Environ Sci Pollut Res Int. 2016 Dec;23(23):23339-23348. doi: 10.1007/s11356-016-7728-4. Epub 2016 Sep 26. PMID 27672044
- [Background] Sun J, Yu G, Zhang Y, Liu X, Du C, Wang L, Li Z, Wang C. Heavy Metal Level in Human Semen with Different Fertility: a Meta-Analysis. Biol Trace Elem Res. 2017 Mar;176(1):27-36. doi: 10.1007/s12011-016-0804-2. Epub 2016 Jul 22. PMID 27444304
- [Background] Le Moal J, Rolland M, Goria S, Wagner V, De Crouy-Chanel P, Rigou A, De Mouzon J, Royere D. Semen quality trends in French regions are consistent with a global change in environmental exposure. Reproduction. 2014 Mar 8;147(4):567-74. doi: 10.1530/REP-13-0499. Print 2014. PMID 24567426
- [Background] Montano L, et al. 2014. Andrology 2(Suppl.2):69, 2014
- [Background] Montano L, et al. 2015. Reprod Toxicol.,Vol. 56: 20,2
- [Background] Bergamo P, Volpe MG, Lorenzetti S, Mantovani A, Notari T, Cocca E, Cerullo S, Di Stasio M, Cerino P, Montano L. Human semen as an early, sensitive biomarker of highly polluted living environment in healthy men: A pilot biomonitoring study on trace elements in blood and semen and their relationship with sperm quality and RedOx status. Reprod Toxicol. 2016 Dec;66:1-9. doi: 10.1016/j.reprotox.2016.07.018. Epub 2016 Sep 1. PMID 27592743
- [Background] Minguez-Alarcon L, Mendiola J, Roca M, Lopez-Espin JJ, Guillen JJ, Moreno JM, Moreno-Grau S, Martinez-Garcia MJ, Vergara-Juarez N, Elvira-Rendueles B, Garcia-Sanchez A, Ten J, Bernabeu R, Torres-Cantero AM. Correlations between Different Heavy Metals in Diverse Body Fluids: Studies of Human Semen Quality. Adv Urol. 2012;2012:420893. doi: 10.1155/2012/420893. Epub 2012 Jan 24. PMID 22312326
- [Background] Zhou N, Cui Z, Yang S, Han X, Chen G, Zhou Z, Zhai C, Ma M, Li L, Cai M, Li Y, Ao L, Shu W, Liu J, Cao J. Air pollution and decreased semen quality: a comparative study of Chongqing urban and rural areas. Environ Pollut. 2014 Apr;187:145-52. doi: 10.1016/j.envpol.2013.12.030. Epub 2014 Feb 1. PMID 24491300
- [Background] Nordkap L, Joensen UN, Blomberg Jensen M, Jorgensen N. Regional differences and temporal trends in male reproductive health disorders: semen quality may be a sensitive marker of environmental exposures. Mol Cell Endocrinol. 2012 May 22;355(2):221-30. doi: 10.1016/j.mce.2011.05.048. Epub 2011 Nov 25. PMID 22138051
- [Background] Verze P, Cai T, Lorenzetti S. The role of the prostate in male fertility, health and disease. Nat Rev Urol. 2016 Jul;13(7):379-86. doi: 10.1038/nrurol.2016.89. Epub 2016 Jun 1. PMID 27245504
- [Background] Eisenberg ML, Li S, Behr B, Pera RR, Cullen MR. Relationship between semen production and medical comorbidity. Fertil Steril. 2015 Jan;103(1):66-71. doi: 10.1016/j.fertnstert.2014.10.017. Epub 2014 Dec 10. PMID 25497466
- [Background] Eisenberg ML, Li S, Behr B, Cullen MR, Galusha D, Lamb DJ, Lipshultz LI. Semen quality, infertility and mortality in the USA. Hum Reprod. 2014 Jul;29(7):1567-74. doi: 10.1093/humrep/deu106. Epub 2014 May 15. PMID 24838701
- [Background] Alegria-Torres JA, Baccarelli A, Bollati V. Epigenetics and lifestyle. Epigenomics. 2011 Jun;3(3):267-77. doi: 10.2217/epi.11.22. PMID 22122337
- [Background] Pacchierotti F, Spano M. Environmental Impact on DNA Methylation in the Germline: State of the Art and Gaps of Knowledge. Biomed Res Int. 2015;2015:123484. doi: 10.1155/2015/123484. Epub 2015 Aug 3. PMID 26339587
- [Background] Cutillas-Tolin A, Minguez-Alarcon L, Mendiola J, Lopez-Espin JJ, Jorgensen N, Navarrete-Munoz EM, Torres-Cantero AM, Chavarro JE. Mediterranean and western dietary patterns are related to markers of testicular function among healthy men. Hum Reprod. 2015 Dec;30(12):2945-55. doi: 10.1093/humrep/dev236. Epub 2015 Sep 25. PMID 26409012
- [Background] Lemyre L, Lalande-Markon MP. Psychological Stress Measure (PSM-9): integration of an evidence-based approach to assessment, monitoring, and evaluation of stress in physical therapy practice. Physiother Theory Pract. 2009 Jul;25(5-6):453-62. doi: 10.1080/09593980902886321. PMID 19842868
- [Background] Riboli E, Kaaks R. The EPIC Project: rationale and study design. European Prospective Investigation into Cancer and Nutrition. Int J Epidemiol. 1997;26 Suppl 1:S6-14. doi: 10.1093/ije/26.suppl_1.s6. PMID 9126529
- [Background] Estruch R, Martinez-Gonzalez MA, Corella D, Salas-Salvado J, Ruiz-Gutierrez V, Covas MI, Fiol M, Gomez-Gracia E, Lopez-Sabater MC, Vinyoles E, Aros F, Conde M, Lahoz C, Lapetra J, Saez G, Ros E; PREDIMED Study Investigators. Effects of a Mediterranean-style diet on cardiovascular risk factors: a randomized trial. Ann Intern Med. 2006 Jul 4;145(1):1-11. doi: 10.7326/0003-4819-145-1-200607040-00004. PMID 16818923
- [Background] Hagstromer M, Oja P, Sjostrom M. The International Physical Activity Questionnaire (IPAQ): a study of concurrent and construct validity. Public Health Nutr. 2006 Sep;9(6):755-62. doi: 10.1079/phn2005898. PMID 16925881
- [Background] Egner PA, Chen JG, Zarth AT, Ng DK, Wang JB, Kensler KH, Jacobson LP, Munoz A, Johnson JL, Groopman JD, Fahey JW, Talalay P, Zhu J, Chen TY, Qian GS, Carmella SG, Hecht SS, Kensler TW. Rapid and sustainable detoxication of airborne pollutants by broccoli sprout beverage: results of a randomized clinical trial in China. Cancer Prev Res (Phila). 2014 Aug;7(8):813-823. doi: 10.1158/1940-6207.CAPR-14-0103. Epub 2014 Jun 9. PMID 24913818
- [Background] Lorenzetti S, Marcoccia D, Mantovani A. Biomarkers of effect in endocrine disruption: how to link a functional assay to an adverse outcome pathway. Ann Ist Super Sanita. 2015;51(2):167-71. doi: 10.4415/ANN_15_02_16. PMID 26156189
- See also: project website — http://www.ecofoodfertility.it/il-progetto/progetto-faast